CLINICAL TRIAL: NCT00334763
Title: Phase II Study of Radiation Followed by Paclitaxel, Carboplatin, and Bevacizumab (PCA) in Patients With Stage IIIB and IV Squamous Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy, Chemotherapy, and Bevacizumab in Treating Patients With Recurrent, Unresectable or Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator felt risk to patients was too high.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Jyoti D. Patel, Robert H. Lurie Comprehensive Cancer Center at Northwestern University
Masking: None | Purpose: Treatment
Other Study IDs: NU 05L1; NU-05L1; NU-1362-038; GENENTECH-AVF3646s
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Biological: bevacizumab
Drug: carboplatin
Drug: chemoprotection
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving radiation therapy together with chemotherapy and monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with chemotherapy and bevacizumab works in treating patients with recurrent, unresectable or stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate reduction in toxicity, in terms of pulmonary hemorrhage, in patients with recurrent, unresectable or stage IIIB or IV squamous non-small cell lung cancer treated with radiotherapy followed by paclitaxel, carboplatin, and bevacizumab.

Secondary

* Determine the overall and progression-free survival of patients treated with this regimen.

OUTLINE: Patients undergo radiotherapy to the primary tumor, clinically involved lymph nodes, and any other disease-causing symptoms or bronchial compression once daily, 5 days a week, for 2 weeks in weeks 1 and 2. Beginning in week 4, patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment with paclitaxel, carboplatin, and bevacizumab repeats every 3 weeks for 4 courses in the absence of unacceptable toxicity. Patients achieving complete response, partial response, or stable disease after 4 courses receive bevacizumab alone as above in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Predominantly squamous cell histology
  * Cytologic or histologic elements can be established on metastatic tumor aspirates or biopsy
* Advanced disease, meeting 1 of the following staging criteria:

  * Stage IIIB disease with malignant pleural effusion
  * Stage IV disease
  * Recurrent, unresectable disease
* Measurable or nonmeasurable disease
* No extrathoracic only disease
* No known CNS metastases by head CT scan with contrast or MRI

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Platelet count > 100,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Bilirubin < 1.5 mg/dL
* Transaminases < 5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 45 mL/min
* Urine protein:creatinine ratio ≤ 1.0 by spot urinalysis
* INR < 1.5 ULN
* PTT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients use effective contraception
* No serious nonhealing wound, ulcer, or bone fracture
* No ongoing or active infection
* No ongoing fever
* No myocardial infarction within the past 6 months
* No stroke within the past 6 months
* No history of hypertension unless well-controlled (i.e., blood pressure < 150/100 mmHg on a stable regimen of antihypertensive therapy)
* No New York Heart Association grade III or IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No unstable angina pectoris
* No peripheral vascular disease ≥ grade 2
* No other clinically significant cardiovascular disease
* No abdominal fistula
* No gastrointestinal perforation
* No intra-abdominal abscess within the past 6 months
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy curatively treated within the past 5 years
* No history of thrombotic or hemorrhagic disorders
* No gross hemoptysis (i.e., red blood ≥ ½ teaspoon) within the past 3 months
* No bleeding requiring intervention or ≥ grade 2

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* No prior systemic chemotherapy for metastatic NSCLC
* More than 6 months since prior adjuvant chemotherapy for early stage (i.e., stage IB-IIIA) NSCLC
* More than 3 weeks since prior immunotherapy, hormonal therapy, or radiotherapy
* More than 28 days since prior and no concurrent major surgery
* More than 7 days since prior minor surgery, fine-needle aspiration, or core biopsy
* More than 4 weeks since prior and no concurrent participation in another experimental drug study
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation of venous access device allowed
* No concurrent chronic treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory drugs known to inhibit platelet function
* No concurrent dipyridamole, ticlopidine, clopidogrel, or cilostazol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Reduction in toxicity measured by pulmonary hemorrhage rate

SECONDARY OUTCOMES:
Overall survival by Kaplan-Meier
Response rate
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti D. Patel, Principal Investigator — Robert H. Lurie Cancer Center
Locations (5):
- United States (5):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas